CLINICAL TRIAL: NCT03951194
Title: Investigating Improvement of Ovarian Function Following Autologous PRP Intra-ovarian Infusion in Perimenopausal Women
Brief Title: Autologous Platelet Rich Plasma (PRP) Intra Ovarian Infusion in Perimenopausal Women
Acronym: PRP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genesis Athens Clinic (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRP- Perimenopause
Record Dates: First submitted 2017-10-25; First posted 2019-05-15 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-01

CONDITIONS: Infertility, Female; Perimenopausal Disorder; Menstrual Cycle Abnormal
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving PRP treatment (Experimental): Perimenopausal women, 40-50 years of age, treated with autologous PRP intra ovarian infusion.
  Interventions: Biological: Autologous Platelet Rich Plasma (PRP) intra ovarian infusion
- Participants receiving Platelet Free Plasma (PFP) (Placebo Comparator): Perimenopausal women, 40-50 years of age, treated with autologous PRP intra ovarian infusion.
  Interventions: Other: Placebo: Autologous Platelet Free Plasma (PFP) intra ovarian infusion

INTERVENTIONS:
Biological: Autologous Platelet Rich Plasma (PRP) intra ovarian infusion — Autologous PRP intra ovarian infusion
  Other Names: PRP; Platelet Rich Plasma
  Arms: Participants receiving PRP treatment
Other: Placebo: Autologous Platelet Free Plasma (PFP) intra ovarian infusion — Autologous PFP intra ovarian infusion
  Other Names: PFP; Platelet Free Plasma
  Arms: Participants receiving Platelet Free Plasma (PFP)

SUMMARY:
Autologous PRP intra ovarian infusion may improve ovarian response and women's hormonal profile and may promote folliculogenesis in perimenopausal women.

DETAILED DESCRIPTION:
This triple-blind Randomized Controlled Trial (RCT) aims to investigate the effectiveness of autologous PRP intra ovarian infusion on improving ovarian tissue functionality and hormonal profile of perimenopausal women. PRP is blood plasma prepared from fresh whole blood that has been enriched with platelets. It is collected from peripheral veins and contains several growth factors such as vascular endothelial growth factor (VEGF), epidermal growth factor (EGF), platelet derived growth factor (PDGF), transforming growth factor (TGF) and other cytokines all of which stimulate tissue proliferation and growth. PRP has been employed in several medical conditions in Orthopedics, Dermatology, and Ophthalmology for wound healing. It's efficacy in ovarian rejuvenation and reactivation and endometrial regeneration has not been fully elucidated. This study aims to investigate the effect of autologous PRP intra ovarian infusion on improving ovarian tissue functionality in perimenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥40 years of age, presenting with cycle irregularities while fulfilling at least one of the respective two criteria: more than seven days difference in menstrual cycle duration between two consecutive cycles OR, presence of a menstrual cycle duration over sixty days and progressive elevation of FSH levels.
* Discontinuation of any complementary/adjuvant treatment including hormone replacement, acupuncture, and botanotherapy, for at least three months prior to recruitment.
* Willing to comply with study requirements

Exclusion Criteria:

* Any pathological disorder related to reproductive system anatomy
* Amenorrhea
* Endometriosis
* Adenomyosis
* Fibroids and adhesions
* Infections in reproductive system
* Current or previous diagnosis of cancer in reproductive system
* History of familiar cancer in reproductive system
* Severe male factor infertility
* Prior referral for PGT
* Ovarian inaccessibility
* Previous POI diagnosis -Endocrinological disorders (Hypothalamus-
* Pituitary disorders, thyroid dysfunction, diabetes mellitus, metabolic syndrome)
* BMI>30 kg/m2 or BMI<18.5 kg/m2
* Systematic autoimmune disorders

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Restoration of menstrual cycle regularity | Three months
  Regular Menstrual cycle
Serum FSH levels | Follow-up period of three months entailing monthly evaluation
  Serum FSH levels evaluated monthly for three consecutive months.

SECONDARY OUTCOMES:
Serum AMH levels | Follow-up period of three months entailing monthly evaluation
  Serum AMH levels evaluated monthly for three consecutive months.
Serum LH levels | Follow-up period of three months entailing monthly evaluation
  Serum LH levels evaluated monthly for three consecutive months.
Serum Estradiol levels | Follow-up period of three months entailing monthly evaluation
  Serum etsradiol levels evaluated monthly for three consecutive months.
Serum Progesteron levels | Follow-up period of three months entailing monthly evaluation
  Serum progesterone levels evaluated monthly for three consecutive months.
Antral Follicle Count | Follow-up period of three months entailing monthly evaluation
  AFC evaluated monthly, on day 2 of the menstrual cycle, for three consecutive months.

CONTACTS AND LOCATIONS:
Overall Officials: Agni Pantou, MD, Study Director — Obstetrician Gynecologist
Locations (1):
- Genesis AC, Athens, Greece